CLINICAL TRIAL: NCT03683342
Title: Comparison of Analgesic Duration of Popliteal Block Versus Ankle Block in Patients Undergoing Forefoot Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Eric Albrecht, Program director of regional anesthesia, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: CER-VD 2018-01090
Record Dates: First submitted 2018-09-20; First posted 2018-09-25 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ankle Block (Active Comparator): Ankle block will be performed under ultrasound guidance.
  Interventions: Procedure: Ankle Block
- Popliteal sciatic nerve block (PSNB) (Active Comparator): PSNB will be performed under ultrasound guidance, along with a saphenous nerve block at the ankle
  Interventions: Procedure: Sciatic nerve block

INTERVENTIONS:
Procedure: Ankle Block — Ankle block will be performed prior to surgery under ultrasound guidance
  Arms: Ankle Block
Procedure: Sciatic nerve block — Sciatic nerve block will be performed prior to surgery under ultrasound guidance
  Arms: Popliteal sciatic nerve block (PSNB)

SUMMARY:
Pain after forefoot surgery can be important and regional anesthesia plays a crucial role in post-operative pain control. Several techniques can be used to achieve surgical anesthesia as well as postoperative analgesia. Of those techniques the ankle block and sciatic nerve block at the popliteal fossa are the most common. The primary goal of this study is thus to compare the analgesic duration of these two types of blocks for patients undergoing forefoot surgery.

DETAILED DESCRIPTION:
Patients scheduled for unilateral forefoot surgery, aged over 18 years old and ASA status I-III without any contra-indications for regional anesthesia will be enrolled.

After a standard randomisation, patients will be allocated in either of two groups : ankle block or sciatic nerve block at the popliteal fossa. In both groups the patients will have a multimodal analgesic regimen followed by a patient-controlled-analgesia (PCA) of morphine.

The primary endpoint is the analgesic duration, defined by the time between the end of the block procedure and the first IV request of morphine from a PCA.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are going to undergo a unilateral forefoot surgery ;
* ASA I-III ;
* Aged 18 years or more;
* Weighing at least 45 kg

Exclusion Criteria:

* Patient refusal and/or language/cognitive barrier
* Pregnancy
* Contra-indication for regional anesthesia
* Opiate or alcohol dependency
* Concomitant oncological disease with chemotherapy
* Patients suffering from neuropathic pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Duration of analgesia | 24 hours after surgery
  Time elapsed between block procedure and first iv request of morphine from PCA

SECONDARY OUTCOMES:
Total opioid consumption at 24h postoperatively | 24 hours after surgery
  Total consumption of morphine from PCA at 24 postoperative hours
Pain score at rest at 4 postoperative hours | 4 hours after surgery
  Pain score (visual analog scale, 0 = minimum; 10 = maximum)
Pain score on movement at 4 postoperative hours | 4 hours after surgery
  Pain score (visual analog scale, 0 = minimum; 10 = maximum)
Pain score at rest at 12 postoperative hours | 12 hours after surgery
  Pain score (visual analog scale, 0 = minimum; 10 = maximum)
Pain score on movement at 12 postoperative hours | 12 hours after surgery
  Pain score (visual analog scale, 0 = minimum; 10 = maximum)
Pain score at rest at 24 postoperative hours | 24 hours after surgery
  Pain score (visual analog scale, 0 = minimum; 10 = maximum)
Pain score on movement at 24 postoperative hours | 24 hours after surgery
  Pain score (visual analog scale, 0 = minimum; 10 = maximum)
Block success rate | 45 minutes after block procedure
  Success of block assessed by pinprick test
Global patient satisfaction 48h after surgery | 48 hours after surgery
  Patient satisfaction score (visual analog scale, 0 = minimum; 10 = maximum)
Complications after block | 48 hours after surgery
  Report of any intravascular injection or any sensory/motor anomalies
Rate of neuropathic pain | 4-6 weeks postoperatively
  Rate of patients describing neuropathic pain 4-6 weeks postoperatively
Rate of paresthesia | Up to 24 hours after block procedure
  Rate of patients complaining of paresthesia
Block procedure time | Up to 10 minutes after ultrasound scanning
  Time from first ultrasound image to needle withdrawal

CONTACTS AND LOCATIONS:
Overall Officials: Eric Albrecht, PD Dr, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- Centre Hospitalier Universitaire Vaudois and University of Lausanne, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Olofsson M, Nguyen A, Rossel JB, Albrecht E. Duration of analgesia after forefoot surgery compared between an ankle and a sciatic nerve block at the popliteal crease: A randomised controlled single-blinded trial. Eur J Anaesthesiol. 2024 Jan 1;41(1):55-60. doi: 10.1097/EJA.0000000000001929. Epub 2023 Nov 16. PMID 37972929